CLINICAL TRIAL: NCT05752266
Title: Effect of Probiotics on Amino Acid Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Technology (Other)
Collaborators: AMILI Pte. Ltd. (Unknown)
Responsible Party: Principal Investigator, Verena Tan Ming Hui, Associate Professor, Singapore Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022180
Record Dates: First submitted 2023-02-17; First posted 2023-03-02 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Protein Digestion; Gastrointestinal Microbiome

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, crossover trial
Who Masked: Participant, Care Provider
Masking Description: Masked personnel will be unaware of which arm each participant is allocated to, and what type of probiotics have been assigned to each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Arm (Experimental): Participants allocated to PRO arm will be administered personalized probiotic pills.
  Interventions: Dietary Supplement: AMILI Probiotic pills
- Placebo Arm (Placebo Comparator): Participants allocated to PRO arm will be administered maltodextrin placebo pills similar in appearance to probiotic pills.
  Interventions: Dietary Supplement: Placebo pills

INTERVENTIONS:
Dietary Supplement: AMILI Probiotic pills — AMILI (AMILI Pte Ltd) will analyze stool samples provided by participants, and assign each participant a type of probiotic pill from the 5 different types of probiotic pills commercially available in AMILI retail store.
  Arms: Probiotic Arm
Dietary Supplement: Placebo pills — Placebo pills contaning maltodextrin with similar appearance to Probiotic pills will be provided to participants allocated to the Placebo Arm.
  Arms: Placebo Arm

SUMMARY:
The goal of this clinical trial is to test effects of consuming probiotics in healthy adults. The main question it aims to answer is:

• Do consuming probiotics affect a healthy adult's ability to absorb amino acids from plant proteins?

Participants will

* Consume one dose of probiotic pills per day after meals for two weeks
* Consume one dose of plant-based plant protein beverage after an overnight fast and collection of one 5 ml fasting blood sample
* Undergo blood draw of 6 more 5 ml blood samples for the next 3 hours after consuming plant-based protein beverage

DETAILED DESCRIPTION:
There is increasing evidence that the gut microbiota contributes to a range of immune, inflammatory, and metabolic responses. Numerous studies have shown that administrating probiotics - strains of bacteria that benefits intestinal function - confer benefits to the host's immune system. Except for soy protein, plant proteins are incomplete proteins lacking in one or more essential amino acids. The incomplete amino acid profile of most plant proteins is compounded by their lower rate of absorption as compared to animal protein. Hence, the investigators aim to investigate the administration of probiotics as a potential strategy to overcome compositional shortcomings of plant proteins by improving the gastrointestinal absorption of plant-based proteins.

The aim of Stage 1 is to formulate a plant-based protein beverage with optimized amino acid profile with consumer acceptance.

Stage 2 of this study will be to conduct a randomized, double-blind, placebo-controlled, crossover trial using the formulation developed in Stage 1, together with probiotics supplementation to evaluate the effect of probiotics on the absorption of amino acids from plant proteins.

The probiotics to be studied will be provided by the Asian Microbiome Library (AMILI) with the plant protein beverage to be developed within SIT. Findings from this mutually beneficial collaborative project with AMILI will pave the way to further understand the role of probiotics in human health, particularly its effect in nutrient absorption of plant protein.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to comply with study procedures and give written informed consent
* Self-reported to be healthy
* Within healthy BMI weight range (18.5-23kg/m2)

Exclusion Criteria:

* Any chronic medical condition
* Individuals who were treated for or diagnosed with a gastrointestinal, cardiac, respiratory, circulatory, musculoskeletal, metabolic, immune, autoimmune, haematological, neurological or endocrinological disorder
* Antibiotic use
* Prebiotics, probiotics, synbiotics, and/or digestive enzymes use
* Food allergy/intolerances/avoidances towards eggs, soya, peanuts, tree nuts, crustaceans, and gluten
* Smoking
* Alcohol consumption

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in blood amino acid concentration | 0 to 150 minutes after ingestion of plant protein beverage on each study visit
  Following ingestion of plant protein beverage, participants will be subjected to drawing of serial blood samples after consuming the plant protein beverage.
  These blood samples will be analyzed for amino acid profile using mass spectrometry methods.
Change in gut microbiota type | 0 to 6 weeks after start of study
  Paricipants will provide a stool sample on each study visit (3 stool samples in total throughout the study). These stool samples given will be analyzed for any changes in type and population size of gut microbes of participants after probiotic intervention and placebo comparator intervention.
Change in gut microbiota population size | 0 to 6 weeks after start of study
  Paricipants will provide a stool sample on each study visit (3 stool samples in total throughout the study). These stool samples given will be analyzed for any changes in type and population size of gut microbes of participants after probiotic intervention and placebo comparator intervention.

SECONDARY OUTCOMES:
Change in blood glucose level | 0 to 150 minutes after ingestion of plant protein beverage
  Following ingestion of plant protein beverage, participants will be subjected to drawing of serial blood samples after consuming the plant protein beverage.
  Serial blood samples will be analyzed for glucose profile using mass spectrometry methods.
Change in blood insulin level | 0 to 150 minutes after ingestion of plant protein beverage
  Following ingestion of plant protein beverage, participants will be subjected to drawing of serial blood samples after consuming the plant protein beverage.
  Serial blood samples will be analyzed for insulin profile using mass spectrometry methods.

CONTACTS AND LOCATIONS:
Overall Officials: Verena Tan, M.Nutr.Diet, Principal Investigator — +65 9172 4062
Locations (1):
- Verena Tan, Singapore, Sinagpore, Singapore

REFERENCES:
- [Background] Jager R, Zaragoza J, Purpura M, Iametti S, Marengo M, Tinsley GM, Anzalone AJ, Oliver JM, Fiore W, Biffi A, Urbina S, Taylor L. Probiotic Administration Increases Amino Acid Absorption from Plant Protein: a Placebo-Controlled, Randomized, Double-Blind, Multicenter, Crossover Study. Probiotics Antimicrob Proteins. 2020 Dec;12(4):1330-1339. doi: 10.1007/s12602-020-09656-5. PMID 32358640

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT05752266/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT05752266/ICF_001.pdf